CLINICAL TRIAL: NCT03233178
Title: Measurement of Alanine Aminotransaminase (ALT) Following Initiation of Antidiabetic Agents in Patients With Type 2 Diabetes in a Real-world Clinical Setting: a Retrospective Cohort Study
Acronym: ALT
Status: Completed | Type: Observational
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: ALT
Record Dates: First submitted 2017-07-20; First posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: T2DM (Type 2 Diabetes Mellitus); Fatty Liver; NAFLD
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fatty Liver; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- SGLT2: Patients initiating SGLT2 inhibitors
  Interventions: Other: Non-interventional
- Liraglutide: Patients initiation liraglutide
  Interventions: Other: Non-interventional
- Sitagliptin: Patients initiating sitagliptin
  Interventions: Other: Non-interventional
- Control Group: Patients who did not initiate any new anti-hyperglycemic treatment
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional

SUMMARY:
The primary objective of this study is to investigate the change in Alanine Aminotransaminase (ALT) in patients with Type 2 Diabetes Mellitus (T2DM) initiating Sodium Glucose Cotransporter 2 (SGLT2) inhibitors, liraglutide, or sitagliptin, compared to a control group of patients who did not initiate a new antihyperglycemic therapy. The hypothesis is that patients using Sodium Glucose Cotransporter 2 inhibitors (SGLT2i) will achieve a greater reduction in ALT compared to the control group.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is very commonly associated with type 2 diabetes mellitus (T2DM) 1. Alanine aminotransferase (ALT) is a common biomarker used to predict levels of NAFLD. The only class of antidiabetic agents thought to be protective of NAFLD are thiazolidinedione's. Few studies have investigated the effect of other antidiabetic agents on bio markers of fatty liver disease 2. A recent pooled analysis of randomized controlled trials that compared canagliflozin to either placebo or sitagliptin showed significant reductions in ALT in the canagliflozin cohorts, which were fully explained by HbA1c and body weight reductions 3. As well, a study that compared ALT change in patients initiating liraglutide found significant reductions in ALT, which was strongly correlated to reduction in body weight 4. However, the effect of different antidiabetic agents on bio markers of fatty liver disease is not well characterized.

The primary objective of this study is to investigate the change in ALT in patients with T2DM initiating SGLT2 inhibitors, liraglutide, or sitagliptin, compared to a control group of patients who did not initiate a new antihyperglycemic therapy. The hypothesis is that patients using SGLT2i will achieve a greater reduction in ALT compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM based upon historical clinical diagnosis
* Patients who initiated canagliflozin, dapagliflozin, liraglutide or sitagliptin by an LMC physician between January 2011 and December 2015, or patients who did not initiate a new diabetes therapy between June 2014 and June 2015.

Exclusion Criteria:

* Diagnosis of type 1 diabetes
* Patients who switched to one of the study treatments from another medication of the same medication class

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include patients with T2DM who are patients at LMC Diabetes & Endocrinology. Patients will be included in the treatment cohorts if they initiated canagliflozin, dapagliflozin, liraglutide or sitagliptin, between January 2011 and December 2015, and did not discontinue the treatment prior to 6 weeks of being on the medication. The control group will include patients with T2DM who are patients at LMC Diabetes & Endocrinology, and who did not initiate any new diabetes treatment between June 2014 and June 2015.
Sampling Method: Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in ALT in patients with T2DM initiating SGLT2 inhibitors, Liraglutide or Sitagliptin compared to control | 1 year
  Change in ALT in patients with T2DM initiating SGLT2 inhibitors, Liraglutide or Sitagliptin compared to control

SECONDARY OUTCOMES:
Change in Hemoglobin A1c from baseline to follow-up | 1 year
  Change in HbA1c from baseline to follow-up
Change in Fasting Plasma Glucose from baseline to follow-up | 1 year
  Change in Fasting Plasma Glucose from baseline to follow-up
Change in body weight from baseline to follow-up | 1 year
  Change in body weight from baseline to follow-up
Change in Body Mass Index (BMI) from baseline to follow-up | 1 year
  Change in BMI from baseline to follow-up
Change in Waist Circumference (WC) from baseline to follow-up | 1 year
  Change in WC from baseline to follow-up
Change in triglycerides from baseline to follow-up | 1 year
  Change in triglycerides from baseline to follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- LMC Brampton, Brampton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bajaj HS, Brown RE, Bhullar L, Sohi N, Kalra S, Aronson R. SGLT2 inhibitors and incretin agents: Associations with alanine aminotransferase activity in type 2 diabetes. Diabetes Metab. 2018 Dec;44(6):493-499. doi: 10.1016/j.diabet.2018.08.001. Epub 2018 Aug 24. PMID 30149145